CLINICAL TRIAL: NCT00556543
Title: Clinical Evaluation of the U-plate Fracture Repair System for the Fixation of Rib Fractures
Brief Title: Clinical Study of the U-Plate Fracture Repair System to Treat Rib Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: ACUTE Innovations, LLC (Industry)
Responsible Party: John Mayberry, MD, Oregon Health & Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 579; eIRB00000579
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Results first posted 2011-05-10 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Rib Fracture; Flail Chest
Keywords: Rib Fracture; Rib Fracture Repair; Rib Fracture ORIF; Flail Chest; Implant; Prosthesis; Rib fracture non-union; Chest wall deformity
MeSH Terms: conditions — Rib Fractures; Flail Chest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Other)
  Interventions: Device: U-plate fracture repair system

INTERVENTIONS:
Device: U-plate fracture repair system — All subjects meeting inclusion criteria will undergo surgery for the repair of their fractured rib/s using the U-plate device. Subjects will be monitored daily during the entire course of their hospitalization for adverse experiences. Subjects will be contacted by phone to complete the MPQ and SF-36 Health Survey. Subjects will be asked if and when they have returned to work or to their previous level of functioning. Subjects will be asked if they had any complications or problems associated with their surgery.

SUMMARY:
The purpose of this study is to gather information about a device used to help fix broken ribs.

Hypothesis: Rib fracture repair with the U-plate system is clinically durable and safe for the indications of flail chest repair, acute pain control, chest wall defect repair, and rib fracture non-union.

DETAILED DESCRIPTION:
Rib fractures are a painful and disabling injury commonly found among trauma patients. According to the National Center for Health Statistics, approximately 300,000 people with rib fractures were treated in emergency and ambulatory care departments in the United States in the year 2004. Rib fracture patients are significantly more disabled at 30 days post-injury than patients with chronic medical illness and lose an average of 70 days of work or usual activity during their acute recovery.

The rationale for conducting this study is to demonstrate in a prospective study that the U-plate repair system is durable and safe. Although this clinical outcome data is not required by the FDA to market and implant this prosthesis, the investigators believe that in order for the U-plate to be widely accepted, prospectively collected outcome data are necessary.

With the goal of improving the durability of fixation of rib fractures over the techniques currently available and with the additional goal of developing a minimally invasive technique, a U-shaped plate was developed. The design of the U-plate theoretically overcomes the inherent softness of the human rib by grasping the rib over its superior margin and by securing the plate with anterior to posterior locking screws that do not rely on screw purchase in bone. Thus much of the strength and durability of the fixation is transferred from the relatively soft rib to the plate itself.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age
* Subjects must have one of the four clinical indications listed below:

  1. Flail chest with failure to wean from ventilator (> 5 days post-injury) and Paradoxical chest wall movement visualized; no significant pulmonary contusion and no significant brain injury
  2. Painful, displaced rib fractures (acute pain control) and failure of narcotics or epidural pain catheter to control pain; fracture movement exacerbates pain (after 7 - 10 days) and minimal associated injuries
  3. Chest wall defect/severely displaced fractures and non-repair defect may result in pulmonary hernia and severely displaced fractures are significantly impeding lung expansion in hemi-thorax
  4. Symptomatic rib fracture non-union and CT scan evidence of fracture non-union at least 2 months post-injury

Exclusion Criteria:

* Subjects who are enrolled in another investigational treatment trial
* Subjects who have received an investigational drug or device within 30 days of enrollment
* Subjects who are unable to complete the follow-up questionnaires
* Subjects with severe head injuries or other severe associated injuries
* Subjects who are not expected to survive the follow-up period
* Female subjects who are pregnant
* Non-English or English as Second Language speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C. Mayberry, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Cacchione RN, Richardson JD, Seligson D. Painful nonunion of multiple rib fractures managed by operative stabilization. J Trauma. 2000 Feb;48(2):319-21. doi: 10.1097/00005373-200002000-00023. No abstract available. PMID 10697096
- [Background] Beal SL, Oreskovich MR. Long-term disability associated with flail chest injury. Am J Surg. 1985 Sep;150(3):324-6. doi: 10.1016/0002-9610(85)90071-6. PMID 4037191
- [Background] Tanaka H, Yukioka T, Yamaguti Y, Shimizu S, Goto H, Matsuda H, Shimazaki S. Surgical stabilization of internal pneumatic stabilization? A prospective randomized study of management of severe flail chest patients. J Trauma. 2002 Apr;52(4):727-32; discussion 732. doi: 10.1097/00005373-200204000-00020. PMID 11956391
- [Background] Ng AB, Giannoudis PV, Bismil Q, Hinsche AF, Smith RM. Operative stabilisation of painful non-united multiple rib fractures. Injury. 2001 Oct;32(8):637-9. doi: 10.1016/s0020-1383(01)00017-1. No abstract available. PMID 11587704

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 Study subjects were enrolled to the study over a 10 month period in 2007 (February to November and underwent surgical repair of their rib fracture injury. All subjects were recruited from the OHSU Hospital and Outpatient Clinic.Study approval was granted on 11/18/2006 by the OHSU Research Integrity Office.
Pre-assignment Details: 6 of the consented study participants had acute rib fractures, 4 had chronic rib fracture non-unions.
Period: Overall Study
Arm/Group | All Study Subjects
Started | 10
Completed | 10 (Subjects completed 180 days of study enrollment)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Subjects
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 46.5 (22.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Rib Fracture [Number; unit: Participants] — Acute Rib Fracture: Subjects with 1. multiple rib fractures and flail chest injury with failure to wean from ventilator (>5 days post-injury, 2. painful, displaced rib fractures who do not receive adequate pain control from usual care, and 3. chest wall defect (visible deformity) / severely displaced rib fractures will be included. Subjects who have sustained a severe head injury or those with extensive associated injuries will not be included.
  Chronic Rib Fracture Non-Union: Subjects with CT evidence of non-healed rib fractures > 2 months from time of injury, with rib pain.
  Participants
    Rib Fracture, Acute | 6
    Rib Fracture, Chronic Non-Union | 4

OUTCOME MEASURES:

1. Primary Outcome: Adverse Post-op Events Related to the Repair and Plating System
Description: Clinical evaluations or chest radiographs at a minimum of 1 and 6 months
Time Frame: 180 days
Population: Per Protocol
Measure: Number; unit: Participants
Groups:
- Acute Rib Fracture Repair: These 6 patients with acute injury underwent rib fracture repair a median of 11 days (range 4 - 18 days) post-injury.
- Rib Fracture Repair for Persistent Rib Fracture Non-Union: Subjects had CT scan evidence of rib fracture non-union at least 3 months from injury date. Subjects were a median of 41.5 months (range 9 - 56 months) post-injury at the time of repair.
Arm/Group | Acute Rib Fracture Repair | Rib Fracture Repair for Persistent Rib Fracture Non-Union
Number analyzed (Participants) | 6 | 4
Participants | 1 | 3
Statistical Analysis 1: Comparison: Acute Rib Fracture Repair vs Rib Fracture Repair for Persistent Rib Fracture Non-Union; Fisher's Exact Test with the null hypothesis that the proportion with adverse events was the same in both groups; Test type: Non-Inferiority or Equivalence — No power calculation performed; p = 0.190, Fisher Exact

2. Primary Outcome: The Rand 36-Item Health Survey Results - Physical Functioning Scale
Description: The RAND 36-Item Short Form Health Survey measures physical and mental health. Study subjects completed the questionnaire at 2 month intervals for 6 months to evaluate net change over time. All questions are scored on a scale from 0 to 100, with 100 representing the highest level of functioning. Aggregate scores are compiled as a percentage of the total points possible, using a RAND scoring table. This health survey was developed at Rand Health as part of the Medical Outcomes Study.
Time Frame: results at 60, 120, and 180 days post-repair with results posted for 180 days
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: RAND-36 scale units
Arm/Group | All Study Subjects
Number analyzed (Participants) | 10
RAND-36 scale units | 65.6 (22.8)

3. Primary Outcome: The Rand 36-Item Health Survey Results - Role Limitations - Physical Scale
Description: as for outcome 2
Time Frame: results at 60, 120, and 180 days post-repair with results posted for 180 days
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: RAND-36 scale units
Arm/Group | All Study Subjects
Number analyzed (Participants) | 10
RAND-36 scale units | 33.3 (35.4)

4. Primary Outcome: The Rand 36-Item Health Survey Results - Role Limitations - Emotional Scale
Description: as for outcome 2
Time Frame: results at 60, 120, and 180 days post-repair with results posted for 180 days
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: RAND-36 scale units
Arm/Group | All Study Subjects
Number analyzed (Participants) | 10
RAND-36 scale units | 81.4 (37.7)

5. Primary Outcome: The Rand 36-Item Health Survey Results - Vitality Scale
Description: as for outcome 2
Time Frame: results at 60, 120, and 180 days post-repair with results posted for 180 days
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: RAND-36 scale units
Arm/Group | All Study Subjects
Number analyzed (Participants) | 10
RAND-36 scale units | 57.2 (18.9)

6. Primary Outcome: The Rand 36-Item Health Survey Results - Emotional Well-being Scale
Description: as for outcome 2
Time Frame: results at 60, 120, and 180 days post-repair with results posted for 180 days
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: RAND-36 scale units
Arm/Group | All Study Subjects
Number analyzed (Participants) | 10
RAND-36 scale units | 73.3 (13.1)

7. Primary Outcome: The Rand 36-Item Health Survey Results - Social Functioning Scale
Description: as for outcome 2
Time Frame: results at 60, 120, and 180 days post-repair with results posted for 180 days
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: RAND-36 scale units
Arm/Group | All Study Subjects
Number analyzed (Participants) | 10
RAND-36 scale units | 76.4 (25.3)

8. Primary Outcome: The Rand 36-Item Health Survey Results - Bodily Pain Scale
Description: as for outcome 2
Time Frame: results at 60, 120, and 180 days post-repair with results posted for 180 days
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: RAND-36 scale units
Arm/Group | All Study Subjects
Number analyzed (Participants) | 10
RAND-36 scale units | 66.0 (24.4)

9. Primary Outcome: The Rand 36-Item Health Survey Results - General Health Scale
Description: as for outcome 2
Time Frame: results at 60, 120, and 180 days post-repair with results posted for 180 days
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: RAND-36 scale units
Arm/Group | All Study Subjects
Number analyzed (Participants) | 10
RAND-36 scale units | 62.2 (20.8)

10. Primary Outcome: The McGill Pain Questionnaire (MPQ) - Present Pain Intensity (PPI)
Description: The MPQ evaluates subjective pain using word descriptors (PPI, present pain intensity) and an intensity scale (PRI, pain rating index). The rank value for each word descriptor is based on its position in the word set. The sum of the rank values is the pain rating index (PPI). The maximum pain score using word descriptors is 78, with a higher score reflecting greater pain.
Time Frame: results at 60, 120, and 180 days post-repair with results posted for 180 days
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: PPI
Arm/Group | All Study Subjects
Number analyzed (Participants) | 10
PPI | 1.22 (0.97)

11. Primary Outcome: The McGill Pain Questionnaire (MPQ) - Pain Rating Index (PRI)
Description: as for outcome 10
Time Frame: results at 60, 120, and 180 days post-repair with results posted for 180 days
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: PRI
Arm/Group | All Study Subjects
Number analyzed (Participants) | 10
PRI | 17.78 (15.58)

ADVERSE EVENTS:
Time Frame: Enrolled subjects were followed for 6 months following surgical repair of their rib fracture.
Description: Subjects were evaluated with radiographic evaluations (chest x-rays) at a minimum of 1 and 6 months. Subjects completed the McGill Pain Questionnaire and the Rand 36 Health Survey at serial intervals during the 6 months of study participation.
Arm/Group | Acute Rib Fracture Repair | Chronic Rib Fracture Non-union Repair
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 1/6 | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Acute Rib Fracture Repair (N=6) | Chronic Rib Fracture Non-union Repair (N=4)
Acute repair adverse event (Infections and infestations) | 1 (1) | 0/0 (0) — There was 1 acute surgical site infection requiring surgical drainage that did not involve the plates. No plating system events occurred in acute fracture repairs.
Chronic non-union repair (Surgical and medical procedures) | 0/0 (0) | 1 (1) — Subject with minimal screw backout on imaging. The subject was asymptomatic and did not require reoperation.
Chronic non-union repair (Surgical and medical procedures) | 0/0 (0) | 1 (1) — Subject experienced complete backout of one screw. The subject was asymptomatic and did not require reoperation.
Chronic non-union repair (Surgical and medical procedures) | 0/0 (0) | 1 (1) — Subject experienced breakage of one metal plate. Plate failure was determined with a chest x-ray. The subject was asymptomatic and did not require reoperation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No